CLINICAL TRIAL: NCT03761511
Title: A Randomized, Double-blind, Placebo-controlled, Parallel-group, Multicentre Study of the Efficacy and Safety of Nicotinamide in Patients With Friedreich Ataxia
Brief Title: Study of the Efficacy and Safety of Nicotinamide in Patients With Friedreich Ataxia
Acronym: NICOFA
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Due to a temporary halt the recruitment start was delayed. A re-evaluation of the sponsor revealed, that the study is no longer feasible due to increased administrative and financial requirements.
Sponsor: RWTH Aachen University (Other)
Collaborators: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 15-138
Record Dates: First submitted 2018-11-27; First posted 2018-12-03 (Actual); Last update posted 2024-01-24 (Actual); Status verified 2024-01

CONDITIONS: Friedreich Ataxia
Keywords: Friedreich Ataxia; Nicotinamide; Rare disease; ZSEA; SARA
MeSH Terms: conditions — Friedreich Ataxia; Rare Diseases | interventions — Niacinamide

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Treatment arm (Active Comparator): Nicotinamide 4 g (capsules) or highest tolerated dose with a minimum of 2 g/d per os once daily
  Interventions: Drug: Nicotinamide
- Placebo arm (Placebo Comparator): Matching Placebo (capsules) once daily
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Nicotinamide — Nicotinamide 4 g (capsules) or highest tolerated dose with a minimum of 2 g/d per os once daily
  Arms: Treatment arm
Drug: Placebo — Matching Placebo (capsules) once daily
  Arms: Placebo arm

SUMMARY:
Friedreich ataxia is the most frequent early-onset autosomal recessive hereditary ataxia. It is caused by a pathological expansion of a GAA repeat in the first intron of the frataxin gene (FXN) and results in decreased levels of FXN protein. FXN deficiency results in a relentlessly progressive neurodegenerative condition which frequently presents around puberty. Patients gradually lose coordination, become dysarthric and are frequently wheel-chair bound as adolescents. There is no disease modifying therapy and many patients die prematurely of cardiomyopathy. It was subsequently found that the FXN gene is silenced at the chromatin level by the formation of heterochromatin and that this heterochromatin formation can be antagonized by histone deacetylase inhibitors (HDACi) (Chan et al., 2013). A recent proof-of-concept clinical study on ten patients with Friedreich ataxia demonstrated that FXN levels can be restored to those seen in asymptomatic carriers using the class III HDACi nicotinamide at a dose that is well tolerated by patients (Libri et al., 2014). Since carriers are asymptomatic, this degree of restoration of FXN expression might be expected to halt disease progression. Nicotinamide readily crosses the blood brain barrier and has previously been given at high doses for long periods to normal individuals without serious adverse effects (Gale et al., 2004; Knip et al., 2000). This study will be the first to provide clinical evidence for the efficacy and safety of nicotinamide in patients with Friedreich´s ataxia.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have a molecular genetic diagnosis of Friedreich ataxia with a GAA- repeat expansion on both alleles of the FXN gene and a SARA Score >7 and <28 and age <50 years.
* Patients must be ≥18 years old and have a weight of at least 50kg.
* Written informed consent prior to study participation
* A female subject is eligible to participate if she is of: Non-childbearing potential defined as pre-menopausal females with a documented tubal ligation or hysterectomy; or postmenopausal defined as 12 months of spontaneous amenorrhea or of childbearing potential and agrees to

Exclusion Criteria:

* Patients with any medical condition or illness that, in the opinion of the investigator would interfere with study compliance and/or impair the patient´s ability to participate or complete the study.
* Any uncontrolled medical or neurological/neurodegenerative condition (other than Friedreich ataxia).
* Clinically significant psychiatric illness (e.g., uncontrolled major depression, schizophrenia, bipolar affective disorder) within 6 months prior to screening.
* Patients with significant clinical dysphagia.
* Hypersensitivity to nicotinamide.
* Patients known to be positive for human immunodeficiency virus (HIV).
* Patients with a significant history of substance abuse (e.g. alcohol or drug abuse) within the previous six months before enrolment.
* Patients with a history of severe allergies to medications.
* Indication of impaired liver function as shown by an abnormal liver function profile at screening (e.g., repeated values of aspartate aminotransferase [AST], alanine aminotransferase [ALT] and bilirubin ≥3 × the upper limit of normal).
* History of malignancy or carcinoma. The following exceptions may be made after discussion with the Sponsor:

  * Subjects with cancers in remission more than 5 years prior to screening.
  * Subjects with a history of excised or treated basal cell or squamous carcinoma.
  * Subjects with prostate cancer in situ.
* History or evidence of an autoimmune disorder considered clinically significant by the Investigator or requiring chronic use of systemic corticosteroids or other immunosuppressants.
* The subject has a history of any other illness, which, in the opinion of the Investigator, might pose an unacceptable risk by administering study medication.
* History of clinically significant cardiac disease (ejection fraction < 40% [normal range 50-70%], cardiac insufficiency defined as New York Heart Association [NYHA] Class >2; clinically significant congenital or acquired valvular disease; symptomatic coronary disease such as prior myocardial infarction or angina, B-type natriuretic peptide (BNP) level increase more than 2 x of the normal age- and gender dependent range; history of unstable arrhythmias, history of atrial fibrillation).
* The subject received an investigational drug within 30 days prior to inclusion into this study.
* Patients taking sodium valproate, tranylcypromine or any other known histone deacetylase inhibitor.
* Use of vitamin B1 (thiamine), withdrawal should be at least 3 months prior screening or 5 half-lives, whichever is longer.
* Use of vitamin B3 (nicotinamide), withdrawal should be at least 3 months prior screening.
* If patients are taking idebenone or coenzyme Q10 (CoQ), this should be stable over the last three months and not changed during the study.
* The subject is unwilling or unable to provide written informed consent and to follow the procedures outlined in the protocol.
* For subjects who will undergo an MRI: Any contraindications to MRI such as, but not limited to cardiac pacemaker, implanted cardiac defibrillator, aneurysm clips, carotid artery vascular clamp, neurostimulator, implanted drug infusion devices, metal fragments or foreign objects in the eyes, skin or body, bone growth/fusion stimulator, cochlear, otologic implant, severe claustrophobia or any condition that would counterindicate an MRI scan.
* Patients participating at start or have been within 30 days before start of study in another pharmacological and non-pharmacological clinical trial, excluding natural history / observational studies.
* The subject is mentally or legally incapacitated.
* Pregnant females as determined by positive [serum or urine] hCG test at Screening or prior to dosing. Participants of child-bearing age should use adequate contraception as defined in the study protocol.
* Lactating females.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2023-04 (Estimated); Primary Completion 2025-06 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Scale for the Assessment and Rating of Ataxia (SARA) | 1 year
  The primary objective of the study is to evaluate the efficacy of daily doses of nicotinamide in slowing disease progression as measured by changes in the Scale for the Assessment and Rating of Ataxia (SARA) as compared with placebo in patients with Friedreich ataxia.
  The SARA is a tool for assessing ataxia. It has eight categories with accumulative score ranging from 0 (no ataxia) to 40 (most severe ataxia). When completing the outcome measure each category is assessed and scored accordingly. Scores for the eight items range as follows:
  Gait (0-8 points), Stance (0-6 points), Sitting (0-4 points) Speech disturbance (0-6 points) Finger chase (0-4 points) Nose-finger test (0-4 points) Fast alternating hand movement (0-4 points) Heel-shin slide (0-4 points) Once each of the 8 categories have been assessed, the total is calculated to determine the severity of ataxia.

SECONDARY OUTCOMES:
Progression of quality of life measures via questionnaire EuroQol five dimensions questionnaire (EQ-5D) | 1 year
  This is a generic instrument, developed and validated by the EuroQoL Group (1990), in which the patient self-rates in particular his/her health status on a visual analogue scale (VAS); the best score is 100.
Modified Friedreich Ataxia Rating Scale (mFARS) | 1 year
  Modified FARS scores are defined as the sum of scores for bulbar function, upper limb coordination, lower limb coordination, and upright stability. The mFARS consists of three subscales, comprising a general score for ataxia, a score for activities of daily living and a neurological examination. The scores can be added to make a total score ranging from 0 to 159. A higher score indicates a greater level of disability.
Progression of cerebellar severity measured by 'Composite Cerebellar Functional Severity´ (CCFS) score | 1 year
  CCFS includes two tests performed with the dominant hand,named the click test and the 9 holes pegboard test (9HPT). An electronic device was created to perform CCFS and to calculate the Z score by subtracting the expected time
Clinician's Global Impression-Change Scale (CGI-C) including comparison of change to the last visit | 1 year
  The Clinical Global Impression - Improvement scale (CGI-I) is a 7 point scale that requires the clinician to assess how much the patient's illness has improved or worsened relative to a baseline state at the beginning of the intervention. and rated as: 1. Very much improved; 2. Much improved; 3. Minimally improved; 4. No change; 5. Minimally worse; 6. Much worse; 7. Very much worse
Safety issues measured by appearance of AEs/SAEs | 1 year
  AEs may be volunteered spontaneously by the patient, or discovered as a result of general non-directed questioning by the study personnel or by physical examination.

CONTACTS AND LOCATIONS:
Locations (7):
- Medical University Innsbruck, Innsbruck, Austria
- Service de génétique médicale - Hôpital La Pitié Salpetrière, Paris, France
- University Hospital RWTH Aachen, Aachen, Germany
- Fondazione IRCCS Istituto Neurologico Carlo Besta, Milan, Italy
- Hospital Universitario La Paz, Madrid, Spain
- United Kingdom (2):
  - Imperial College London, London
  - University College London, London

IPD SHARING:
Plan to Share IPD: Undecided
The study results will be published in appropriate international scientific journals, and publishing details will be given in the clinical study agreement. The study will be registered and study results will be disclosed by the principal investigator in one or more public clinical study registry(ies), according to national/international use.

REFERENCES:
- [Derived] Reetz K, Hilgers RD, Isfort S, Dohmen M, Didszun C, Fedosov K, Kistermann J, Mariotti C, Durr A, Boesch S, Klopstock T, Rodriguez de Rivera Garrido FJ, Schols L, Klockgether T, Pandolfo M, Korinthenberg R, Lavin P, Molenberghs G, Libri V, Giunti P, Festenstein R, Schulz JB; EFACTS or NICOFA study group. Protocol of a randomized, double-blind, placebo-controlled, parallel-group, multicentre study of the efficacy and safety of nicotinamide in patients with Friedreich ataxia (NICOFA). Neurol Res Pract. 2019 Oct 15;1:33. doi: 10.1186/s42466-019-0038-9. eCollection 2019. PMID 33324899
- Available data/document: Study Protocol: NICOFA — https://ukaachen.sharepoint.com/:b:/s/NICOFA/ESUAT8h1fTBHlTcsdu48LrQBbvvAABdsy81bvQ4Egq696g?e=8Xliis

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-12-05): https://cdn.clinicaltrials.gov/large-docs/11/NCT03761511/Prot_SAP_000.pdf